CLINICAL TRIAL: NCT03907930
Title: Comparative Study Between Tubeless and Standard Percutaneous Nephrolithotomy. Randomized Controlled Trial (RCT)
Brief Title: Conventional PCNL Versus Tubeless PCNL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Alsayed Ahmed Zowita, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: tubeless PCNL
Record Dates: First submitted 2019-03-28; First posted 2019-04-09 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Percutaneous Nephrolithotomy

STUDY DESIGN:
Intervention Model Description: group of patients will be submitted for conventional PCNL other group will be submitted to tubeless PCNL
Who Masked: Participant, Care Provider, Investigator
Masking Description: triple blinded study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional (Active Comparator): this arm will have both nephrostomy tube and ureteric catheter after completing the operation
  Interventions: Procedure: percutaneous nephrolithotripsy
- tubeless (Active Comparator): the arm will have only ureteric catheter rafter completing the operation
  Interventions: Procedure: percutaneous nephrolithotripsy

INTERVENTIONS:
Procedure: percutaneous nephrolithotripsy — removal of kidney and upper ureteric stones through small incision in the loin using nephroscope after disintegration by lithoclast
  Other Names: PCNL

SUMMARY:
prospective randomized study measuring the safety and efficacy of tubeless PNL in patients at assiut university hospital comparing to the standard PNL

DETAILED DESCRIPTION:
Percutaneous nephrolithotomy (PNL) is considered to be the procedure of choice for the treatment of upper urinary tract calculi. It was first introduced in 1976, and since that the operative technique and the endoscopic equipments underwent many modifications to increase the success rates and to decrease complications.

Because of high success rate, low morbidity and complication rate, this minimally invasive modality has replaced the open surgical approach. the standard procedure is to place nephrostomy tubes within the tract of varying caliber and types.

This was done to facilitate maximal collecting system drainage, to tamponade the access tract and also securing the access in case of 2nd look PNL was needed. multiple studies demonstrate significant morbidity associated with nephrostomy tube following PNL, mainly postoperative pain that requires significant narcotic and also long hospital stay. the idea of the "tubeless" PCNL was born, whereby a nephrostomy tube is not left in place following the percutaneous procedure, but rather renal drainage is established with an indwelling ureteral stent. Tubeless PNL has been challenged by certain problems as regard the selection of the patients. Another problem that is facing the tubeless PNL may be is the question regarding the access tract and how to deal with?. Finally, Percutaneous nephrolithotomy (PCNL) has become the standard treatment for kidney stones and/or upper ureter, but Whether nephrostomy tube placement is necessary after PCNL is still a matter of debate

ELIGIBILITY:
Inclusion Criteria:

* Patients above 18 years old 2. Patients with any stone burden and stone number requiring single procedure

Exclusion Criteria:

1 - Patients aged below 18 years old. 2. Anatomical variation of the kidney in shape or position, e.g. horseshoe kidney or malrotation.

3. Complex or staghorn stones requiring staged procedure.

Intra operative criteria:

4. Three or more access tracts. 5. Significant intraoperative bleeding. 6. Intraoperative pelvi calyceal system perforation. 7. Residual stones necessitate 2nd look PNL

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-03-28 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
number of days of hospital stay for both groups | 15 days
  comparison between number of days in hospital for both groups
dose of analgesia used to control pain after the procedure | 5 days
  comparison between the dose of analgesia needed for both groups in milligram

CONTACTS AND LOCATIONS:
Overall Officials: atef abd aziz, professor, Study Chair — assuit university hospital urology departement egypt
Locations (1):
- Assuit University Hospitals, Asyut, Egypt

REFERENCES:
- [Background] Fernstrom I, Johansson B. Percutaneous pyelolithotomy. A new extraction technique. Scand J Urol Nephrol. 1976;10(3):257-9. doi: 10.1080/21681805.1976.11882084. PMID 1006190
- [Background] Valdivia Uria JG, Valle Gerhold J, Lopez Lopez JA, Villarroya Rodriguez S, Ambroj Navarro C, Ramirez Fabian M, Rodriguez Bazalo JM, Sanchez Elipe MA. Technique and complications of percutaneous nephroscopy: experience with 557 patients in the supine position. J Urol. 1998 Dec;160(6 Pt 1):1975-8. doi: 10.1016/s0022-5347(01)62217-1. PMID 9817303